CLINICAL TRIAL: NCT00212810
Title: TOPAMAX (Topiramate) Intervention to Prevent Transformation of Episodic Migraine: The Topiramate INTREPID Study
Brief Title: Evaluation of the Effectiveness of Topiramate in Preventing the Transformation From Episodic Migraine to Chronic Daily Headache.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002854
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Migraine; Headache; Classic Migraine; Common Migraine
Keywords: Migraine; Headache; Migraine Headache
MeSH Terms: conditions — Migraine Disorders; Headache; Migraine with Aura; Migraine without Aura | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to determine whether Topiramate is effective in preventing the development of chronic daily headache among patients with episodic migraine headaches.

DETAILED DESCRIPTION:
Chronic daily headache encompasses a frequent headache state in which the increased burden of pain further compromises quality of life and adversely impacts patients, their families, and health care providers. Approximately 5% of patients with migraine, or an estimated 1.4 million Americans, manifest a chronic daily headache form of disease. The consequences include resistance to treatment, worsening quality of life, increased use and over use of medication, and development of ischemic and other neuropathological brain lesions. This is a randomized, double-blind, placebo-controlled multicenter study that will enroll patients 18-65 years old with an established history of migraine headaches who, in the 28 days prior to the study should have a migraine frequency of at least 10 but less than 15 migraine headache days per month, and less than 15 total headache days (migraine plus non migraine headaches) per month. The study duration will be approximately 26 weeks. The study is divided into 4 phases as follows: A Screening/Washout Phase that may last between 2-6 weeks, depending on whether you need to stop taking a medication that is not allowed in the study; A Baseline Phase lasting 4 weeks, at which time information will be collected on the migraine and non-migraine headaches you experience during this period; A double-blind Titration Phase lasting 4-6 weeks where all patients will be randomized to treatment with either Topiramate or placebo. If you are randomized to Topiramate, your dose will be gradually increased up to a dose of either 75 or 100 mg a day; A Maintenance Period lasting 20 weeks at which time you will continue on the dose you were taking at the completion of the Titration period; and a Taper/Exit phase, lasting 2 weeks, where you will gradually reduce the dose of study medication you were taking during the study. The study hypothesis is that the study drug will be more effective than placebo in preventing patients from transforming from episodic migraines to chronic daily headaches. Each patient will be asked to record their headache pain information and medication use on paper headache diaries. Patients will receive either Topiramate or placebo. The number of tablets of topiramate or placebo, will be gradually increased to either a minimum of 3 tablets/day or a maximum of 4 tablets/day. For those on Topiramate, 3 tablets would represent 75 mg and 4 tablets would represent 100 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* To qualify for this study you must be 18-65 years old
* have a history of migraine headaches for at least 1 year
* experience at least 10 but less than 15 migraine headache days and less than 15 total headache days/month
* able to take oral medication
* able to understand and sign the informed consent and to complete headache diaries.

Exclusion Criteria:

* You will not be able to participate in the study if you previously discontinued Topiramate because it did not make you feel better or it made you feel different
* have migraine aura without headache
* have a positive urine drug screen
* have a history of kidney stones
* have a history of suicide attempt
* pregnant females
* already on a migraine preventive medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2005-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter will be whether or not a patient experiences 15 or more headache days (migraine and non-migraine) during the last 28 days of the study.

SECONDARY OUTCOMES:
Time to development of transformed migraine;occurrence of transformation as function of baseline headache days;change in the average rate of migraine days;percentage change in the average rate of migraine days;50%,75%, and 100% reduction in migraine days

CONTACTS AND LOCATIONS:
Overall Officials: Ortho McNeil Neurologics, Inc. Clinical Trial, Study Director — Ortho-McNeil Neurologics, Inc.

REFERENCES:
- [Derived] Lipton RB, Silberstein S, Dodick D, Cady R, Freitag F, Mathew N, Biondi DM, Ascher S, Olson WH, Hulihan J. Topiramate intervention to prevent transformation of episodic migraine: the topiramate INTREPID study. Cephalalgia. 2011 Jan;31(1):18-30. doi: 10.1177/0333102410372427. Epub 2010 May 17. PMID 20974598
- See also: The Topiramate INTREPID Study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=917&filename=CR002854_CSR.pdf